CLINICAL TRIAL: NCT01812772
Title: The Effect of Ureteric Stent Tethers on Patient Symptoms, Stent Bacterial Colonization and Urinary Tract Infection
Brief Title: The Effect of Ureteric Stent Tethers on Patient Symptoms and Urinary Infection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-370
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2014-02

CONDITIONS: Kidney Stone
Keywords: urinary stents; ureteroscopy
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Double J-stent with a long tether (Experimental): Following ureteroscopy patients will have placed a double J-stent with a long tether.
  Interventions: Device: Double J-stent with a long tether
- Double J-stent without a long tether (Active Comparator): Following ureteroscopy patients will have a double J-stent placed without a long tether
  Interventions: Device: Double J-stent without a long tether

INTERVENTIONS:
Device: Double J-stent with a long tether — Patients will receive a double-J stent placement with a long tether following ureteroscopy.
  Arms: Double J-stent with a long tether
Device: Double J-stent without a long tether — Patients will receive a double-J stent placement without a long tether following ureteroscopy.
  Arms: Double J-stent without a long tether

SUMMARY:
RESEARCH QUESTION Do ureteric stents with tethers, left in-situ for 1-2 weeks, increase the rate of stent bacterial colonization, urinary bacterial colonization and stent related lower urinary tract symptoms compared to stents without tethers?

HYPOTHESIS We hypothesize that ureteral double-J stents with tethers increase the rate of stent bacterial colonization, but do not increase the rate of urinary bacterial colonization or stent related lower urinary tract symptoms compared to stents without tethers when left in-situ for 1-2 weeks.

DETAILED DESCRIPTION:
Two of the main issues surrounding the use of ureteral stents are stent related symptoms and bacterial colonization/urinary tract infection (UTI). To be useful, stent tethers must decrease the morbidity associated with stent removal and the cost to the health care system, while not increasing stent related symptoms or UTI. To our knowledge, the effect of leaving a stent tether on stent symptoms and bacterial colonization of the stent and urine has not been previously studied.

This is a single-centre, prospective, randomized, controlled trial. Patients eligible for recruitment into the study based on the inclusion and exclusion criteria will be provided with a consent form at the time of their initial appointment, when their ureteroscopy is being booked. Once consent is obtained, patients will be randomized (using random number table look-up) to receive either double-J stent placement with a tether (the Treatment Group) or double-J stent placement without a tether (the Control Group) following ureteroscopy. Randomization will occur prior to the commencement of ureteroscopy.

Patients will either have a double J-stent placed with or without a long tether attached. The double-J stents used in the treatment and control groups will be otherwise identical. All stents will be 6 French in diameter and 22-26 cm in length based on the patients' height. Sizing of stent length will be performed uniformly in the treatment and control group and will involve measuring ureteric length from the ureteropelvic junction to ureterovesical junction with a marked ureteral catheter. All patients will receive a single preoperative dose of prophylactic antibiotics (i.e., Ampicillin and Gentamicin or Ciprofloxacin).All patients will have a urine sample collected for culture and sensitivity at the start of the procedure.

Blinding will not be feasible during this trial due to the nature of the intervention. The urologist performing the procedure will clearly be aware of whether a tether is left on the stent. Similarly, patients will also be aware of whether a string tether is protruding from their urethral meatus or not. However, assessors of the compiled data and questionnaires will be blinded to the intervention.

Once enrolled in the study, patients will be given the Ureteral Stent Symptoms Questionnaire 1 (Pre Stent) to complete prior to undergoing ureteroscopy and stent insertion. This will allow us to establish baseline lower urinary tract symptoms.

After completion of ureteroscopy and stent insertion and upon discharge from the hospital all patients will be provided with the following:

1. Diary sheets to record daily analgesic use
2. A prescription for a standardized analgesic regimen including Percocet (1 tablet PO q6h prn, 20 tablets) to be taken as needed for pain control.
3. An appointment for the first follow-up visit (in 7-14 days)

At the follow-up visit, a kidney, ureter and bladder (KUB) radiograph will be performed and patients will complete the Ureteral Stent Symptoms Questionnaire 2 (Stent insitu). The KUB x-ray will be reviewed to ensure the stent remained in appropriate position and did not migrate and that any residual stone fragments have passed. Next, all patients will have their stent removed. Patients in the control group will undergo cystoscopy under local anesthesia for stent removal and those the treatment group will have the stent removed by the tether. This distal curl or lower end (bladder) of the double-J stent, in all patients, will be sent to microbiology for culture to determine the rate of stent bacterial colonization. Of note, all patients in the control group will provide a mid-stream urine sample to be sent for culture and sensitivity testing, after cystoscopy and stent removal, while all patients in the treatment group will provide a urine sample after the stent is removed, so the tether does not contaminate the sample. This urine sample will allow us to establish the rate of bacteriuria.

Upon discharge from the Cystoscopy unit following stent removal all patients will return for a final follow-up with renal ultrasound approximately 4-6 weeks post-stent removal and will be given the Ureteral Stent Symptoms Questionnaire 3 (Post Stent) to complete.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years
2. First presentation for ureteroscopy for this particular stone
3. Planned insertion of a double J-stent
4. Follow-up conducted at St. Michael's Hospital

Exclusion Criteria:

1. Age <18years
2. Preexisting stent in place
3. Bilateral ureteric stents to be inserted
4. Patients with congenital kidney anomalies (horseshoe kidney, ectopic kidney, etc.)
5. Patients with an indwelling foley catheter
6. Patients with neurogenic bladder, chronic prostatitis, painful bladder syndrome or interstitial cystitis
7. Patients with a urinary diversion (ileal conduit, ileal neobladder)
8. Patient currently taking an α-blocker (alfuzosin, terazosin,tamsulosin, prazosin)
9. Active urinary tract infection or positive screening urine culture at preadmission
10. Pregnancy
11. Patients who will not be returning to St. Michael's Hospital for follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The difference in stent related lower urinary tract symptoms based on mean scores from the Ureteral Stent Symptoms questionnaires | The Ureteral Stent Symptoms Questionnaires will be completed before the procedure, 1 week after the procedure and 1 month after the stent was removed (5 weeks post procedure)

SECONDARY OUTCOMES:
the rate of stent bacterial colonization | 1 week post procedure

CONTACTS AND LOCATIONS:
Overall Officials: R. John D Honey, MD FRCSC, Principal Investigator — Unity Health Toronto; Kenneth T Pace, MD FRCSC, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael Hospital, Toronto, Ontario, Canada